CLINICAL TRIAL: NCT02415647
Title: Longitudinal Family/Molecular Genetic Study to Validate Research Domain Criteria
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen V. Faraone, Faculty, State University of New York - Upstate Medical University
Other Study IDs: 543389-8; R01MH101519-01A1 (NIH)
Record Dates: First submitted 2015-03-31; First posted 2015-04-14 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Mental Disorders; Psychological Disorders; Psychiatric, Diagnosis; Mental Disorders Diagnosed in Childhood
Keywords: children; mental health; family genetic study
MeSH Terms: conditions — Mental Disorders; Neurodevelopmental Disorders; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Child Proband with Psychiatric Disorder: Affected group of child probands with psychiatric disorders (ages 6-12 years).
- Normal Comparison Group: Non-disordered psychiatrically normal comparison group (ages 6-12 years).

SUMMARY:
The purpose of this research is to study new ways of classifying mental disorders in children based on observable behavior and genetics to ultimately diagnose these disorders better.

DETAILED DESCRIPTION:
The NIMH Research Domain Criteria (RDoC) initiative seeks to further a long-range goal of contributing to diagnostic systems as informed by research on genetics, neuroscience, and behavior. The RDoC approach is based on identifying the most elemental units of analysis relevant to psychiatric disorders (such as genes and molecules) and using this matrix as a framework for investigation. In this case-control family study, the investigators will be using self-report questionnaires and computer-based tests to develop diagnostic methods for neuropsychiatric disorders in children, their siblings, and their parents. They will do this by recruiting "normal" and "affected" children, their siblings, and their parents. They will look at the subject, sibling, and parents to determine if psychiatric disorders are inherited. "Affected" children, ages 6-12, are those who have been diagnosed with a psychiatric disorder. Participants will undergo a battery of questionnaires/evaluations and a blood draw. The investigators will determine if the questionnaires and tests that reflect the constructs (such as reward prediction and willingness to work) predict psychopathology and impairment. The blood draw will be genotyped to determine if the measured constructs are associated with neuropsychiatric candidate genes, cross-disorder candidate gens and a cross-disorder polygenic score.

ELIGIBILITY:
Inclusion Criteria:

* male or female, ages 6-12.
* biological child of parent(s) participating in testing.

Exclusion Criteria:

* taking psychotropic medications.
* free of uncontrolled medical problems.
* major sensorimotor disability (e.g., deafness, blindness).
* diagnosed neurological condition.
* inadequate command of the English language.
* history of head injury with loss of consciousness lasting longer than 10 minutes.
* IQ estimated at below 80.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Child probands with psychiatric disorders will be recruited from psychiatric clinics, child psychiatrists, and mental health providers in Onondaga County. Non-disordered psychiatrially normal comparison groups will be recruited from a pediatric primary care clinic.
Sampling Method: Probability Sample
Enrollment: 2806 (Actual)
Dates: Start 2014-10; Primary Completion 2018-09-13 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Reward Valuation | Baseline
  Measures: Self-report, computerized tests, and DNA samples; Assessing correlations among family members and predictors of psychopathology.
Effort Valuation/Willingness to Work | Baseline
  Measures: Self-report, computerized tests, and DNA samples; Assessing correlations among family members and predictors of psychopathology.
Expectancy/Reward Prediction Error | Baseline
  Measures: Self-report, computerized tests, and DNA samples; Assessing correlations among family members and predictors of psychopathology.
Initial Responsiveness to Reward Attainment | Baseline
  Measures: Self-report, computerized tests, and DNA samples; Assessing correlations among family members and predictors of psychopathology.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Faraone, Ph.D., Principal Investigator — Upstate Medical University
Locations (1):
- Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Glatt SJ, Stone WS, Faraone SV, Seidman LJ, Tsuang MT. Psychopathology, personality traits and social development of young first-degree relatives of patients with schizophrenia. Br J Psychiatry. 2006 Oct;189:337-45. doi: 10.1192/bjp.bp.105.016998. PMID 17012657
- [Background] Faraone SV, Seidman LJ, Kremen WS, Kennedy D, Makris N, Caviness VS, Goldstein J, Tsuang MT. Structural brain abnormalities among relatives of patients with schizophrenia: implications for linkage studies. Schizophr Res. 2003 Apr 1;60(2-3):125-40. doi: 10.1016/s0920-9964(02)00304-3. PMID 12591577
- [Background] Faraone SV, Su J, Tsuang MT. A genome-wide scan of symptom dimensions in bipolar disorder pedigrees of adult probands. J Affect Disord. 2004 Oct;82 Suppl 1:S71-8. doi: 10.1016/j.jad.2004.05.015. PMID 15571792
- [Background] Glatt SJ, Su JA, Zhu SC, Zhang R, Zhang B, Li J, Yuan X, Li J, Lyons MJ, Faraone SV, Tsuang MT. Genome-wide linkage analysis of heroin dependence in Han Chinese: results from wave one of a multi-stage study. Am J Med Genet B Neuropsychiatr Genet. 2006 Sep 5;141B(6):648-52. doi: 10.1002/ajmg.b.30361. PMID 16856125
- [Background] Glatt SJ, Faraone SV, Lasky-Su JA, Kanazawa T, Hwu HG, Tsuang MT. Family-based association testing strongly implicates DRD2 as a risk gene for schizophrenia in Han Chinese from Taiwan. Mol Psychiatry. 2009 Sep;14(9):885-93. doi: 10.1038/mp.2008.30. Epub 2008 Mar 11. PMID 18332877
- [Background] Cross-Disorder Group of the Psychiatric Genomics Consortium. Identification of risk loci with shared effects on five major psychiatric disorders: a genome-wide analysis. Lancet. 2013 Apr 20;381(9875):1371-1379. doi: 10.1016/S0140-6736(12)62129-1. Epub 2013 Feb 28. PMID 23453885
- [Background] Faraone SV, Matise T, Svrakic D, Pepple J, Malaspina D, Suarez B, Hampe C, Zambuto CT, Schmitt K, Meyer J, Markel P, Lee H, Harkavy Friedman J, Kaufmann C, Cloninger CR, Tsuang MT. Genome scan of European-American schizophrenia pedigrees: results of the NIMH Genetics Initiative and Millennium Consortium. Am J Med Genet. 1998 Jul 10;81(4):290-5. PMID 9674973
- [Background] Faraone SV, Biederman J, Mick E, Wozniak J, Kiely K, Guite J, Ablon JS, Warburton R, Reed E. Attention deficit hyperactivity disorder in a multigenerational pedigree. Biol Psychiatry. 1996 May 15;39(10):906-8. doi: 10.1016/0006-3223(95)00194-8. No abstract available. PMID 8860195
- [Background] Faraone SV, Adamson JJ, Wilens TE, Monuteaux MC, Biederman J. Deriving phenotypes for molecular genetic studies of substance use disorders: a family study approach. Drug Alcohol Depend. 2007 May 11;88(2-3):244-50. doi: 10.1016/j.drugalcdep.2006.11.002. Epub 2006 Dec 1. PMID 17141426
- [Background] Faraone SV, Adamson JJ, Wilens TE, Monuteaux MC, Biederman J. Familial transmission of derived phenotypes for molecular genetic studies of substance use disorders. Drug Alcohol Depend. 2008 Jan 1;92(1-3):100-7. doi: 10.1016/j.drugalcdep.2007.07.002. Epub 2007 Sep 4. PMID 17766060